CLINICAL TRIAL: NCT06128954
Title: A Phase I, Single Centre, Randomised, Interventional, Open-Label, Cross-Over Study to Evaluate the Pharmacokinetics (PK) and the Safety and Tolerability of a Total Daily Dose of 900mg of TETA 4HCL, Comparing a New Once Daily TETA 4HCL Formulation (300mg) (3x300mg Trientine Base Tablets, OD) With the Current Marketed Cuprior® Formulation (150mg) (3x150mg Trientine Base Tablets, BD) in Adult Healthy Male and Female Participants
Brief Title: Study Comparing Once Daily Dose of 900mg of TETA 4HCL Against Cuprior® (450mg Trientine Base, Twice Daily).
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Orphalan (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: ORPH-131-012
Record Dates: First submitted 2023-11-02; First posted 2023-11-13 (Actual); Results first posted 2025-08-15 (Actual); Last update posted 2025-08-15 (Actual); Status verified 2025-08

CONDITIONS: Wilson's Disease
MeSH Terms: conditions — Hepatolenticular Degeneration

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Once Daily Dose Formulation (Treatment A) (Experimental): 1 x 900mg TETA 4HCl, new once daily formulation (3x300mg trientine base tablets as a single AM dose)
  Interventions: Drug: 900mg TETA 4HCl Once Daily Formulation
- Cuprior® comparator (Treatment B) (Active Comparator): 2 x 450mg TETA 4HCl, Marketed Cuprior® formulation (6 x150mg trientine base tablets in two equally divided doses (450mg doses 8 hours apart)
  Interventions: Drug: 900mg TETA 4HCl Cuprior®

INTERVENTIONS:
Drug: 900mg TETA 4HCl Once Daily Formulation — 3x300mg trientine base tablets as a single AM dose
  Arms: Once Daily Dose Formulation (Treatment A)
Drug: 900mg TETA 4HCl Cuprior® — 6 x150mg trientine base tablets in two equally divided doses
  Arms: Cuprior® comparator (Treatment B)

SUMMARY:
A randomised, open-label study evaluating the pharmacokinetics, safety, and tolerability of a new once daily dose of 900mg of TETA 4HCL by comparing it against the current marketed Cuprior® formulation (450mg trientine base, twice daily) in healthy male and female participants.

DETAILED DESCRIPTION:
This is a single centre, phase I, randomized, controlled trial with a crossover design to evaluate the pharmacokinetics (PK), safety, and tolerability of a new once daily TETA 4HCL formulation (300mg) (3x300mg trientine base tablets, OD) compared to the current marketed Cuprior® formulation (150mg) (3x150mg trientine base tablets, BD) in adult healthy male and female participants.

Participants: 26 healthy participants will be enrolled to ensure 24 participants complete the study, with a balanced gender split.

Treatment: Participants will be randomized to receive either the new or the current formulation of the drug, and then switch to the other formulation after a period of time (see study flow chart below).

To remain in line with current EU SmPC and US PIL, being:

* EU daily dose range of 450-975 mg of trientine base
* US daily dose range of 150-1500mg trientine base the following treatments will be administered according to the treatment allocation schedule below: A: 900mg TETA 4HCl once a day / new formulation = 3 tablets of 300mg trientine base as a single dose B: 900mg TETA 4HCl marketed Cuprior formulation = 6 tablets of 150mg trientine base in two equally divided doses

Patients will be randomised in a 1:1 ratio to either one of the following sequences:

Treatment Sequence Period 1 Period 2 Sequence 1 Treatment A Treatment B Sequence 2 Treatment B Treatment A

Assessments: Participants will be assessed for eligibility criteria and will be monitored closely throughout the study. Assessments will be performed during the study and at the end of the study follow-up visit.

Duration: The duration of the study will be up to approximately 7 weeks, from screening to follow-up:

* Screening will take place between days -28 and -2
* In-house period from D-1 to D3 with dosing on D1 of each treatment period
* Follow-up will take place on D7 of Treatment Period 2

At least 5 days and a maximum of 10 days between treatment period study drug administration

Objective: To evaluate the PK, safety, and tolerability of the new once daily TETA 4HCL formulation compared to the current marketed Cuprior® formulation.

ELIGIBILITY:
Inclusion Criteria:

* Age: 18 to 40 years
* Body weight: ≥ 50 kg
* BMI: 18.0 to 25.0 kg/m2
* Health: Generally healthy, with no clinically significant illnesses or surgeries in the past 12 weeks
* Willingness to comply with trial procedures and restrictions

Exclusion Criteria:

* Significant current or recurrent disease
* Acute significant disease or illness within 7 days before the start of the trial
* Clinically significant deviations in blood tests
* An estimated glomerular filtration rate (eGFR) of less than 60 ml/min/1.73m2
* Positive test for alcohol, drugs of abuse, hepatitis B surface antigen (HBsAg), hepatitis C antibody (HCV Ab), or human immunodeficiency virus antibody (HIV Ab)
* Pregnant or breastfeeding women
* History or regular use of tobacco or other nicotine-containing products within 6 months before the start of the trial
* Treatment with an investigational drug within 90 days or 5 half-lives (whichever is longer) or exposure to more than 3 investigational drugs within 12 months of first study drug administration
* Use of prescription medication (excluding female hormonal contraception or hormone replacement therapy)within 30 days or 5 half
* lives (whichever is longer) prior to first study drug administration, or use of over-the-counter (OTC) medication (including multivitamin, herbal, or homeopathic preparations; Paracetamol use ≤2g per day is permitted) during the 14 days or 5 half-lives of the drug (whichever is longer) before first study drug administration
* History of sensitivity/allergy to the study medications or components thereof (mannitol, colloidal anhydrous silica, glycerol dibehenate or magnesium-stearate)
* Donation or loss of 450 mL or more of blood or plasma within 16 weeks prior to first trial medication administration or intention to donate blood in the 16 weeks after completing the trial
* An inability to follow a standardised diet and meal schedule or inability to fast, as required during the trial
* Participants deemed to have difficult veins for cannulation/blood draws

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 26 (Actual)
Dates: Start 2024-01-16 (Actual); Primary Completion 2024-02-08 (Actual); Study Completion 2024-02-16 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Thomas Ashdown, MBBCh Ssc, Principal Investigator — Richmond Pharmacology Limited
Locations (1):
- Richmond Pharmacology Ltd, London, United Kingdom

RESULTS

PARTICIPANT FLOW:
Groups:
- Sequence 1: Once Daily TETA 4HCl Formulation, Followed by Twice Daily Cuprior® Formulation: Participants first received 1 x 900mg TETA 4HCl, once daily formulation (3x300mg trientine base tablets as a single AM dose), for 3 days. After a washout period of a minimum of 5 days and up to 10 days, they then received 2 x 450mg TETA 4HCl, marketed Cuprior® formulation (6 x150mg trientine base tablets in two equally divided doses (450mg doses 8 hours apart) for 3 days.
- Sequence 2: Twice Daily Cuprior® Formulation, Followed by Once Daily TETA 4HCl Formulation: Participants first received 2 x 450mg TETA 4HCl, marketed Cuprior® formulation (6 x150mg trientine base tablets in two equally divided doses (450mg doses 8 hours apart), for 3 days. After a washout period of a minimum of 5 days and up to 10 days, they then received 1 x 900mg TETA 4HCl, once daily formulation (3x300mg trientine base tablets as a single AM dose) for 3 days.
Period: Overall Study
Arm/Group | Sequence 1: Once Daily TETA 4HCl Formulation, Followed by Twice Daily Cuprior® Formulation | Sequence 2: Twice Daily Cuprior® Formulation, Followed by Once Daily TETA 4HCl Formulation
Started | 13 | 13
Completed | 13 | 13
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: Cross over design of two treatment sequences where 26 study participants are studied in both sequences.
Groups:
- Total: Total of all reporting groups
Arm/Group | Sequence 1: Once Daily TETA 4HCl Formulation, Followed by Twice Daily Cuprior® Formulation | Sequence 2: Twice Daily Cuprior® Formulation, Followed by Once Daily TETA 4HCl Formulation | Total
Number analyzed (Participants) | 13 | 13 | 26
Age, Continuous [Mean (Standard Deviation); unit: years] | 26.4 (5.82) | 28.5 (5.91) | 27.4 (5.85)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7 | 6 | 13
  Male | 6 | 7 | 13
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2 | 0 | 2
  Not Hispanic or Latino | 11 | 13 | 24
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 1 | 1 | 2
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 4 | 4
  White | 10 | 5 | 15
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 2 | 3 | 5

OUTCOME MEASURES:

1. Primary Outcome: Plasma Concentrations (AUC) of TETA 4HCL Following Administration of Two TETA 4HCL Tablet Formulations.
Description: PK parameters derived by non-compartmental methods including: AUC 24 and AUCinf. PK sampling was done pre-first dose and then post-first dose for Treatment A (hours): 0.5, 1, 1.25, 1.5, 2, 3, 4, 5, 6, 8, 12, 16, 24, 36, 48. Post-first dose for Treatment B (hours): 0.5, 1, 1.25, 1.5, 2, 3, 4, 5, 6, 8 (before 2nd dose), 8.5, 9, 9.25, 9.5, 10, 11, 12, 13, 14, 16, 20, 24, 36, 48.
Time Frame: Up to 48 hours post first dose initiation.
Measure: Geometric Mean (90% Confidence Interval); unit: h*ng/mL
Arm/Group | Once Daily Dose Formulation (Treatment A) | Cuprior® Comparator (Treatment B)
Number analyzed (Participants) | 26 | 26
h*ng/mL
  AUC 24 | 12668.493 [10236.595 to 15678.135] | 10971.720 [8865.542 to 13578.262]
  AUCinf | 13561.621 [10956.316 to 16786.442] | 11778.232 [9515.532 to 14578.980]

2. Primary Outcome: Plasma Concentrations (AUC) of N1-acetyltriethylenetetramine (MAT) Following Administration of Two TETA 4HCL Tablet Formulations.
Description: as for outcome 1
Time Frame: Up to 48 hours post first dose initiation.
Measure: Geometric Mean (90% Confidence Interval); unit: h*ng/mL
Arm/Group | Once Daily Dose Formulation (Treatment A) | Cuprior® Comparator (Treatment B)
Number analyzed (Participants) | 26 | 26
h*ng/mL
  AUC 24 | 19327.926 [17712.265 to 21090.962] | 25318.882 [23202.426 to 27628.396]
  AUCinf | 23383.874 [21524.239 to 25404.176] | 30655.260 [28217.358 to 33303.790]

3. Primary Outcome: Plasma Concentrations (AUC) of N1, N10-diacetyltriethylenetetramine (DAT) Following Administration of Two TETA 4HCL Tablet Formulations.
Description: as for outcome 1
Time Frame: Up to 48 hours post first dose initiation.
Measure: Geometric Mean (90% Confidence Interval); unit: h*ng/mL
Arm/Group | Once Daily Dose Formulation (Treatment A) | Cuprior® Comparator (Treatment B)
Number analyzed (Participants) | 26 | 26
h*ng/mL
  AUC 24 | 4966.208 [4159.876 to 5928.837] | 6310.627 [5286.009 to 7533.852]
  AUCinf | 6285.164 [5358.373 to 7372.253] | 8324.132 [7096.681 to 9763.883]

4. Primary Outcome: Pharmacokinetic Parameters (AUC) of TETA in Plasma
Description: PK parameters derived by non-compartmental methods including: AUCinf and AUC 24. PK sampling was done pre-first dose and then post-first dose for Treatment A (hours): 0.5, 1, 1.25, 1.5, 2, 3, 4, 5, 6, 8, 12, 16, 24, 36, 48. Post-first dose for Treatment B (hours): 0.5, 1, 1.25, 1.5, 2, 3, 4, 5, 6, 8 (before 2nd dose), 8.5, 9, 9.25, 9.5, 10, 11, 12, 13, 14, 16, 20, 24, 36, 48.
Time Frame: Up to 48 hours post first dose initiation.
Population: Crossover design, participants exposed to both treatments.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: h*ng/mL
Arm/Group | Once Daily Dose Formulation (Treatment A) | Cuprior® Comparator (Treatment B)
Number analyzed (Participants) | 26 | 26
h*ng/mL
  AUCinf | 13561.621 (48.627) | 11778.232 (45.404)
  AUC 24 | 12668.493 (49.498) | 10971.720 (45.807)

5. Primary Outcome: Plasma Concentrations (Cmax) of TETA 4HCL Following Administration of Two TETA 4HCL Tablet Formulations.
Description: PK parameters derived by non-compartmental methods including: Cmax.
Time Frame: Up to 48 hours post first dose initiation.
Measure: Geometric Mean (90% Confidence Interval); unit: ng/mL
Arm/Group | Once Daily Dose Formulation (Treatment A) | Cuprior® Comparator (Treatment B)
Number analyzed (Participants) | 26 | 26
ng/mL | 3435.621 [2876.753 to 4103.061] | 1567.145 [1312.220 to 1871.595]

6. Primary Outcome: Pharmacokinetic Parameters (Time) of TETA in Plasma
Description: PK parameters derived by non-compartmental methods including: Thalf and Tmax.
Time Frame: Up to 48 hours post first dose initiation.
Population: Crossover design, participants exposed to both treatments.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Hours
Arm/Group | Once Daily Dose Formulation (Treatment A) | Cuprior® Comparator (Treatment B)
Number analyzed (Participants) | 26 | 26
Hours
  Thalf | 15.593 (30.461) | 8.643 (49.617)
  Tmax | 0.8874 (73.6544) | 1.9438 (116.0599)

7. Primary Outcome: Pharmacokinetic Parameters (Concentration) of TETA in Plasma
Description: PK parameters derived by non-compartmental methods including: Clast and Cmax.
Time Frame: Up to 48 hours post first dose initiation.
Population: Crossover design, participants exposed to both treatments.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | Once Daily Dose Formulation (Treatment A) | Cuprior® Comparator (Treatment B)
Number analyzed (Participants) | 26 | 26
ng/mL
  Clast | 16.040 (45.710) | 17.382 (44.905)
  Cmax | 3436 (41) | 1567 (45)

8. Primary Outcome: Pharmacokinetic Parameters (AUC) of MAT in Plasma
Description: as for outcome 4
Time Frame: Up to 48 hours post first dose initiation
Population: Crossover design, participants exposed to both treatments.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: h*ng/mL
Arm/Group | Once Daily Dose Formulation (Treatment A) | Cuprior® Comparator (Treatment B)
Number analyzed (Participants) | 26 | 26
h*ng/mL
  AUCinf | 23383.874 (27.676) | 30655.260 (22.052)
  AUC 24 | 19327.926 (29.416) | 25318.882 (22.149)

9. Primary Outcome: Plasma Concentrations (Cmax) of N1-acetyltriethylenetetramine (MAT) Following Administration of Two TETA 4HCL Tablet Formulations.
Description: PK parameters derived by non-compartmental methods including: Cmax.
Time Frame: Up to 48 hours post first dose initiation.
Measure: Geometric Mean (90% Confidence Interval); unit: ng/mL
Arm/Group | Once Daily Dose Formulation (Treatment A) | Cuprior® Comparator (Treatment B)
Number analyzed (Participants) | 26 | 26
ng/mL | 2030.958 [1849.766 to 2229.898] | 2058.668 [1875.003 to 2260.323]

10. Primary Outcome: Pharmacokinetic Parameters (Time) of MAT in Plasma
Description: PK parameters derived by non-compartmental methods including: Thalf and Tmax..
Time Frame: Up to 48 hours post first dose initiation
Population: Crossover design, participants exposed to both treatments.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Hours
Arm/Group | Once Daily Dose Formulation (Treatment A) | Cuprior® Comparator (Treatment B)
Number analyzed (Participants) | 26 | 26
Hours
  Thalf | 13.852 (27.030) | 9.045 (16.633)
  Tmax | 3.8785 (26.4810) | 13.0875 (12.7188)

11. Primary Outcome: Pharmacokinetic Parameters (Concentration) of MAT in Plasma
Description: PK parameters derived by non-compartmental methods including: Clast and Cmax..
Time Frame: Up to 48 hours post first dose initiation
Population: Crossover design, participants exposed to both treatments.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | Once Daily Dose Formulation (Treatment A) | Cuprior® Comparator (Treatment B)
Number analyzed (Participants) | 26 | 26
ng/mL
  Clast | 67.119 (32.127) | 81.886 (36.080)
  Cmax | 2031 (32) | 2059 (23)

12. Primary Outcome: Pharmacokinetic Parameters (AUC) of DAT in Plasma
Description: as for outcome 4
Time Frame: Up to 48 hours post first dose initiation.
Population: Crossover design, participants exposed to both treatments.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: h*ng/mL
Arm/Group | Once Daily Dose Formulation (Treatment A) | Cuprior® Comparator (Treatment B)
Number analyzed (Participants) | 26 | 26
h*ng/mL
  AUCinf | 6285.164 (51.082) | 8324.132 (50.170)
  AUC 24 | 4966.208 (56.026) | 6310.627 (55.882)

13. Primary Outcome: Plasma Concentrations (Cmax) of N1, N10-diacetyltriethylenetetramine (DAT) Following Administration of Two TETA 4HCL Tablet Formulations.
Description: PK parameters derived by non-compartmental methods including: Cmax.
Time Frame: Up to 48 hours post first dose initiation.
Measure: Geometric Mean (90% Confidence Interval); unit: ng/mL
Arm/Group | Once Daily Dose Formulation (Treatment A) | Cuprior® Comparator (Treatment B)
Number analyzed (Participants) | 26 | 26
ng/mL | 443.208 [362.437 to 541.979] | 450.705 [368.568 to 551.147]

14. Primary Outcome: Pharmacokinetic Parameters (Time) of DAT in Plasma
Description: PK parameters derived by non-compartmental methods including: Thalf and Tmax.
Time Frame: Up to 48 hours post first dose initiation.
Population: Crossover design, participants exposed to both treatments.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Hours
Arm/Group | Once Daily Dose Formulation (Treatment A) | Cuprior® Comparator (Treatment B)
Number analyzed (Participants) | 26 | 26
Hours
  Thalf | 11.053 (14.335) | 8.529 (11.086)
  Tmax | 5.3587 (14.9105) | 12.3653 (20.6338)

15. Primary Outcome: Pharmacokinetic Parameters (Concentration) of DAT in Plasma
Description: PK parameters derived by non-compartmental methods including: Clast and Cmax.
Time Frame: Up to 48 hours post first dose initiation.
Population: Crossover design, participants exposed to both treatments.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | Once Daily Dose Formulation (Treatment A) | Cuprior® Comparator (Treatment B)
Number analyzed (Participants) | 26 | 26
ng/mL
  Clast | 22.899 (33.640) | 30.100 (37.799)
  Cmax | 443 (64) | 451 (63)

16. Secondary Outcome: To Compare the Safety and Tolerability of the Two TETA 4HCL Tablet Formulations.
Description: The incidence, severity, and relationship of Treatment-Emergent Adverse Events (TEAEs).
Time Frame: Adverse events were collected from the patient signing the ICF until the end of study/follow-up (EOS/FU) visit. The Mean (Min, Max) number of days between signing ICF and the EOS/FU visit in the study was 20.2 (16, 25). All patients completed the study.
Measure: Count of Participants; unit: Participants
Arm/Group | Once Daily Dose Formulation (Treatment A) | Cuprior® Comparator (Treatment B)
Number analyzed (Participants) | 26 | 26
Participants
  Participants with treatment-related TEAEs. | 2 | 1
  Participants with clinically significant changes in laboratory safety tests | 0 | 0
  Participants with morphological and/or rhythm abnormalities on electrocardiogram (ECG) | 0 | 0
  Participants with clinically significant changes in vital signs | 0 | 1

ADVERSE EVENTS:
Time Frame: Adverse events were collected from the patient signing the ICF until the end of study/follow-up (EOS/FU) visit. The Mean (Min, Max) number of days between signing ICF and the EOS/FU visit in the study was 20.2 (16, 25). All patients completed the study.
Arm/Group | Once Daily Dose Formulation (Treatment A) | Cuprior® Comparator (Treatment B)
All-Cause Mortality (participants affected / at risk) | 0/26 | 0/26
Serious Adverse Events (participants affected / at risk) | 0/26 | 0/26
Other Adverse Events (participants affected / at risk) | 3/26 | 3/26
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Once Daily Dose Formulation (Treatment A) (N=26) | Cuprior® Comparator (Treatment B) (N=26)
Presyncope (Cardiac disorders) | 0 (0) | 1 (1)
Abdominal discomfort (Gastrointestinal disorders) | 0 (0) | 1 (1)
Aphthous ulcer (Gastrointestinal disorders) | 1 (1) | 0 (0)
Epigastric discomfort (Gastrointestinal disorders) | 1 (1) | 0 (0)
Nausea (Gastrointestinal disorders) | 1 (1) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 0 (0) | 1 (1)
Viral infection (Infections and infestations) | 0 (0) | 1 (1)
Rash macular (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Full study agreement in place with Richmond Pharmacology.

DOCUMENTS (3):
  • Study Protocol and Statistical Analysis Plan: Study Protocol (2024-01-09): https://cdn.clinicaltrials.gov/large-docs/54/NCT06128954/Prot_SAP_000.pdf
  • Statistical Analysis Plan: Statistical Analysis Plan (2024-01-31): https://cdn.clinicaltrials.gov/large-docs/54/NCT06128954/SAP_001.pdf
  • Informed Consent Form (2024-01-17): https://cdn.clinicaltrials.gov/large-docs/54/NCT06128954/ICF_002.pdf